CLINICAL TRIAL: NCT01617525
Title: A Comparison of the Effects on Cardiovascular Risk Factors of Korean and American Dietary Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Korean Diet Study
Record Dates: First submitted 2012-03-31; First posted 2012-06-12 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Korean Recommended Diet (Experimental): A dietary pattern that follows the recommendations by the Korean Rural Development Administration.
  Interventions: Other: Controlled Feeding Dietary Intervention
- US Recommended Diet (Active Comparator): Diet based on recipes and menus developed by the USDA Dietary Guidelines for Americans intramural team.
  Interventions: Other: Controlled Feeding Dietary Intervention
- Typical American Diet (Active Comparator): Diet based on data from the NHANES surveys, as summarized in the USDA report What We Eat in America.
  Interventions: Other: Controlled Feeding Dietary Intervention

INTERVENTIONS:
Other: Controlled Feeding Dietary Intervention — All meals will be provided during each 4-week intervention period. Participants must consume all foods provided and must not consume any outside foods during each intervention period.

SUMMARY:
The primary aim of this study is to compare, in a group of at-risk individuals, the role of three dietary patterns on indices of Cardiovascular Disease (CVD) risk: a) the recommended Korean pattern; b) the typical American diet, based on national dietary intake surveys; and c) the 2010 DGA diet pattern. A secondary aim will be to assess the effects of each diet on intestinal microbiota and on inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Non Asian-American men and women between the ages of 25-65 years
* Body Mass Index (BMI) ≥ 25 and ≤ 38 kg/m2
* Fasting LDL-cholesterol ≥ 130 mg/dL
* Willingness and ability to make scheduled appointments at clinical site as required by study protocol

Exclusion Criteria:

* Major aversions to Korean foods
* Known food allergies that would interfere with study protocol
* Use of cholesterol-lowering medication or dietary supplements
* Use of blood pressure medications
* Use of prebiotics or probiotics in the last 3 months
* Received medication for bacterial infection (antibiotic) in the last 3 months
* Regular use of fiber supplements or laxatives
* Conditions requiring ongoing medical care and/or medication, including kidney, liver, gastrointestinal or endocrine disorders.
* Regular tobacco use within 6 months prior to the start of the study
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Voluntary or involuntary weight loss of 10% of body weight within the last 12 months
* Self-report of alcohol or substance abuse within the past 12 months
* Donated blood during the 8 week period prior to the study
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study anticipation or the ability to follow the intervention protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Disease Biomarkers | End of each 4-week diet period
  Plasma total cholesterol, HDL and LDL cholesterol, insulin, glucose, and serum triglycerides will be measured.

SECONDARY OUTCOMES:
Inflammatory Markers | End of each 4-week diet
  Cytokine production will be analyzed by selecting representative pro-inflammatory cytokine genes (i.e. TNF-a, IL-12, IL-6, IFNg), anti-inflammatory genes (IL-10), and different signaling pathways (i.e. Mitogen activated protein kinase (MAPK) p38, phosphatidylinositol 3 (PI3) kinase, and nuclear factor Kappa B (NF-KB).
Markers of appetite and food intake regulation | End of each 4-week diet
  Plasma adiponectin, ghrelin, PYY and leptin will be measured.
Blood pressure | End of each 4-week diet
Urinary sodium excretion, potassium, urea nitrogen, phosphorus, and creatinine | End of each 4-week diet
Change in fecal microbiota | At baseline and after 4-weeks of each diet
  Fecal samples will be collected to study changes in bacterial abundance of commensal microorganisms such as Bifidobacterium spp., Lactobacillus spp., E.coli spp. and Bacteroides fragilis spp.
Dietary Questionnaires | At end of each 4-week diet
  Participants will be asked to complete questionnaires regarding acceptability, satiety, and gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Derived] Schroeder N, Park YH, Kang MS, Kim Y, Ha GK, Kim HR, Yates AA, Caballero B. A randomized trial on the effects of 2010 Dietary Guidelines for Americans and Korean diet patterns on cardiovascular risk factors in overweight and obese adults. J Acad Nutr Diet. 2015 Jul;115(7):1083-92. doi: 10.1016/j.jand.2015.03.023. PMID 26115560